CLINICAL TRIAL: NCT01442571
Title: Hyaluronic Acid Injection Post Arthroscopy - Does it Improve Immediate Function? Double Blind Controlled Prospective Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sports01-CTIL-HMO
Record Dates: First submitted 2011-09-04; First posted 2011-09-28 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-08

CONDITIONS: Cartilage Injury
Keywords: Adult Men and Women, who underwent arthroscopy of the knee with cartilage injury of ICRS grade 2 or higher
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyaluronic Acid Injection, pain, function (Experimental)
  Interventions: Device: Hyaluronic Acid Injection
- Saline Injection (Placebo Comparator)
  Interventions: Drug: Saline Injection

INTERVENTIONS:
Device: Hyaluronic Acid Injection
  Arms: Hyaluronic Acid Injection, pain, function
Drug: Saline Injection
  Arms: Saline Injection

SUMMARY:
The proposed research is to examine the effect of injecting a large volume of HA (10cc) at the time of post arthroscopy suture removal (9-11 day post surgery), in patients with cartilage damage of ICRS grade 2 and above in one of the knee compartments.

ELIGIBILITY:
Inclusion Criteria:

* Adult Men and Women, who underwent arthroscopy of the knee with cartilage injury of ICRS grade 2 or higher in one of the compartments (in addition to other injuries such as meniscal tear and cruciate ligament).

Exclusion Criteria:

* Patients with known rheumatic disorders.
* Known hypersensitivity to HA.
* Synovial diseases like PVNS, under 18y old.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)

PRIMARY OUTCOMES:
IKDC (the International Knee Documentation Committee)

CONTACTS AND LOCATIONS:
Locations (1):
- Jerusalem, Israel